CLINICAL TRIAL: NCT07242742
Title: Effectiveness of Pulpotomy vs. Root Canal Treatment in Extremely Deep Caries: A Randomized Controlled Trial Conducted in Supervised Undergraduate Clinics
Brief Title: Effectiveness of Pulpotomy vs. Root Canal Treatment in Extremely Deep Caries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-4505
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Extremely Deep Caries; Pulpitis
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: care providers and participants are masked at the start of caries removal and up to the stage of random allocation to pulpotomy or root canal treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full Pulpotomy (Experimental): The intra-operative standard care for pulpotomy is as follows:
  * Clinical procedure should be completed over one or 2 visits
  * Performed under local anaesthesia and rubber dam isolation
  * Complete caries removal
  * Pulp resection using sterile high-speed bur with water coolant
  * Irrigation protocol with 1.25% sodium hypochlorite
  * Haemostasis with a 1.25% sodium hypochlorite-moistened cotton pellet over the amputated pulps for up to 10 minutes
  * Placement of Biodentine (Septodont Ltd., Saint Maur des Fausse s, France) or its alternative approved by NUCOHS for pulpotomy
  * Final definitive resin-based restoration
  * Post-operative periapical radiograph taken
  Interventions: Procedure: Full Pulpotomy
- Root Canal Treatment (Active Comparator): The intra-operative standard care for root canal treatment is as follows:
  * Clinical procedure can be carried out over one or 2 visits
  * Use of rubber dam mandatory
  * Irrigation protocol with 1.25% sodium hypochlorite
  * Working length with combined radiographs and apex locators
  * Automated instrumentation to accompany hand instrumentation
  * Preparation to apical size 2-3 larger than largest file that binds at the WL in the uninstrumented canal initial apical file (IAF)
  * Canal medicament; non setting calcium hydroxide if done in two visits
  * Root canal filling with gutta pecha and traditional sealers (cold lateral or warm vertical condensation)
  * Ensure coronal seal
  * Good quality postoperative radiograph using parallel cone technique
  * Final restoration as per undergraduate clinical protocols
  Interventions: Procedure: root canal treatment and intracanal medicament

INTERVENTIONS:
Procedure: Full Pulpotomy — Preservation of vital pulp tissue for tooth survival.
  Arms: Full Pulpotomy
Procedure: root canal treatment and intracanal medicament — Root canal treatment as a comparator to pulpotomy.
  Arms: Root Canal Treatment

SUMMARY:
Recent clinical trials comparing pulpotomy versus root canal treatment (RCT) have shown promising outcomes; however, the current evidence lacks generalisability to general practitioners. It remains to be elucidated whether these favourable results can be replicated in a primary care setting. This study aims to address that gap by involving senior dental students undergoing supervised university education and training, with the potential to inform future best practice guidelines and promote the adoption of vital pulp therapy (VPT) as a predictable treatment alternative in the general dental population.

The clinical procedure involves complete caries-free excavation carried out under rubber dam isolation. After confirming vital pulp status-demonstrated by bleeding upon entry, participants will be randomised to receive one of two treatments: RCT or full pulpotomy.

Outcomes will include clinical and radiographic success or failure of the intervention at 12 months. Additionally, patient-reported outcomes will be collected, specifically pain experienced and the use of analgesia during the immediate post-operative period (days 3 and 7).

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 years or older
* Mature maxillary or mandibular permanent tooth with extremely deep restorations/caries penetrating the entire thickness of dentine on the radiograph without a radiopaque zone separating the lesion from the pulp (Bjorndal et al., 2019)
* Tooth may or may not be symptomatic at the time of recruitment but must be responsive to cold and EPT sensibility testing
* Tooth is restorable and can be adequately isolated during treatment
* One tooth per patient

Exclusion Criteria:

* Teeth with difficult access and unpredictable isolation using a rubber dam
* Teeth aberrant root canal morphology, extreme root curvatures (>30 degrees), calcified canals/sclerosed pulp
* Teeth indicated for elective root canal treatment for restorative purposes
* Teeth with apical periodontitis
* Presence of apical radiolucency
* Any evidence of purulence or excessive bleeding that cannot be controlled with a cotton pellet with 1.25% hypochlorite for 10 minutes
* History of trauma to the tooth
* Teeth with active periodontal disease (pocket depth >5mm)
* Patients with complex medical histories that may affect their caries experience and healing ability (immunocompromised, radiotherapy etc.)
* Patients who are pregnant or breast-feeding
* Patients who are unable to consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 12 months
  Clinical and radiographic success or failure of the intervention will be measured at 12 months. The primary outcome is a composite measure at 12 months: 1) absence of pain indicative of unhealthy pulp; 2) absence of signs and symptoms indicative of acute or chronic periapical disease; 3) absence of radiographic evidence of failure including radiolucency or resorption. Failure of any part of the composite, at or any time before 12 months, will equate to overall treatment failure.

SECONDARY OUTCOMES:
Secondary Outcome | 12 months
  A patient reported outcome of pain experienced and use of analgesia in the immediate post-operative period (days 3, 7) will be collected through a paper questionnaire distributed at visit 1. The presence of a structurally integral tooth with an intact, nondefective restoration at 12 months, with positive sensibility response to EPT and with absence of need for any further intervention during the 12-month follow-up period, presence of calcification or adverse event will be reported on. A parallel health economics analysis will be completed using data collected from participants at baseline and at 12 months using common agreed templates.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Centre For Oral Health Singapore (NUCOHS), Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Only anonymised data can be shared, subject to local health records governance.
Supporting Information: Study Protocol, SAP